CLINICAL TRIAL: NCT01905020
Title: An Open-label, Randomized, Three-way, Multicenter Study to Compare the Efficacy of Single-hormone Closed-loop Strategy, Dual-hormone Closed-loop Strategy and Conventional Insulin Pump Therapy in Regulating Overnight Glucose Levels at Home in Adolescents and Adults With Type 1 Diabetes
Brief Title: Closed-loop Control of Overnight Glucose Levels in Adults and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Montreal Children's Hospital of the MUHC (Other); Mount Sinai Hospital, New York (Other); McGill University (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-04
Record Dates: First submitted 2013-07-12; First posted 2013-07-22 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia; Insulin; Glucagon; Closed-loop system; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional insulin pump therapry (Active Comparator): Subjects will use conventional pump therapy to regulate their glucose levels.
  Interventions: Other: Carbohydrate-rich meal; Other: Exercise
- Single-hormone closed-loop system (Active Comparator): Variable subcutaneous insulin infusion rate will be used to regulate glucose levels. Insulin Aspart (Novorapid) will be infused using a subcutaneous infusion pump. The glucose level as measured by the real time sensor will be entered manually into the computer every 10 minutes. The pump's infusion rate will then be changed manually based on the computer-generated recommendations of infusion rates.
  Interventions: Other: Carbohydrate-rich meal; Other: Exercise
- Dual-hormone closed-loop system (Active Comparator): Insulin Aspart (Novorapid) and glucagon (Paladin) will be infused using two separate subcutaneous infusion pumps. The glucose levels as measured by the real time sensor will be entered manually into the computer every 10 minutes. The pumps' infusion rate will then be changed manually based on the computer generated-recommendation delivery levels.
  Interventions: Other: Carbohydrate-rich meal; Other: Exercise

INTERVENTIONS:
Other: Carbohydrate-rich meal — At 19:30, patients will eat a standardized large meal (110g carbohydrate for males; 90g carbohydrate for females). Conventional insulin pump therapy or closed-loop system will be use to control glucose levels from 21:00 until 7:00 next morning.
Other: Exercise — Study participants will go to a training facility around 18:00 to perform a 60min workout at 60% heart rate reserve. The workout will be on a treadmill and/or a stationary bicycle. Conventional insulin pump therapy or closed-loop system will be use to regulate glucose levels from 21:00 until 7:00 next morning.

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormone: insulin and glucagon.

The main objective of this project is to compare the efficacy of single-hormone closed-loop strategy, dual-hormone closed-loop strategy and pump therapy to regulate overnight glucose levels in a out-patient study in adults and adolescents with type 1 diabetes.

The investigators hypothesized that dual-hormone closed-loop strategy is more effective in regulating overnight glucose levels in adults and adolescents with type 1 diabetes compared to single-hormone closed-loop strategy, which in turn is more effective than the conventional pump therapy.

DETAILED DESCRIPTION:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormone: insulin and glucagon.

We aim to conduct a multicenter study to compare the efficacy of conventional pump therapy, single-hormone closed-loop strategy and dual-hormone closed-loop strategy to regulate overnight glucose levels, at home, in adolescents and adults with type 1 diabetes. Each intervention will be tested on two nights: 1) After a carbohydrate-rich dinner meal (to exaggerate hyperglycemic risk and; 2) After an evening exercise (to exaggerate hypoglycemic risk).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 12 years of old.
* Body mass index < 35
* Clinical diagnosis of type 1 diabetes for at least one year.
* The subject will have been on insulin pump therapy for at least 4 months.
* HbA1c < 12%.
* At least two visits with an endocrinology team in the past 1 year.

Exclusion Criteria:

* Clinically significant nephropathy, neuropathy (peripheral or autonomic e.g. significant gastroparesis) or retinopathy as judged by the investigator.
* Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* A recent injury to body or limb, muscular disorder, use of any medication or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol.
* Ongoing pregnancy.
* Severe hypoglycemic episode within two weeks of screening.
* Current use of glucocorticoid medication (except low stable dose and inhaled therapy).
* Known or suspected allergy to the insulin aspart, glucagon, Medtronic sensors, or Medtronic infusion sets..
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
* Anticipating a significant change in treatment regimen between admissions (such as a major change in an exercise routine, significant change in dietary routine or in insulin therapy.
* Failure to comply with team's recommendations.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percentage of time in target range | 8 hours
  Percentage of time for which glucose levels (as measured by the glucose sensor) are in target range. Target range is defined to be between 4.0 to 8.0 mmol/L

SECONDARY OUTCOMES:
Percentage of time in target range for each night separately | 8 hours
  Percentage of time for which glucose levels are in target range for each night separately. Target range is defined to be between 4.0 and 8.0 mmol/L.
Percentage of time in target range for the pooled data | 8 hours
  Percentage of time for which glucose levels are in target range for the pooled data. Target range is defined to be between 4.0 to 8.0 mmol/L.
Percentage of time spent below 4.0 mmol/L | 8 hours
  Percentage of time for which glucose levels are below 4.0 mmol/L.
Percentage of time spent below 3.3 mmol/L | 8 hours
  Percentage of time for which glucose levels are spent below 3.3 mmol/L.
Area under the curve for glucose levels below 4.0 mmol/L | 8 hours
Area under the curve for glucose levels below 3.3 mmol/L | 8 hours
Percentage of time spent above 8.0 mmol/L | 8 hours
  Percentage of time for which glucose levels are above 8.0 mmol/L
Percentage of time spent above 10.0 mmol/L | 8 hours
  Percentage of time for which glucose levels are above 10.0 mmol/L.
Area under the curve for glucose levels spent above 8.0 mmol/L | 8 hours
Area under the curve for glucose levels spent above 10.0 mmol/L | 8 hours
Mean glucose levels | 8 hours
Standard deviation of glucose levels | 8 hours
  Standard deviation of glucose levels as a measure of glucose variability.
Total insulin delivery | 8 hours
Number of subjects experiencing at least one hypoglycemic event requiring treatment | 8 hours
Number of hypoglycemic events requiring treatment | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal; Bruce Perkins, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Toronto, Ontario
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - Montreal Children Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Haidar A, Rabasa-Lhoret R, Legault L, Lovblom LE, Rakheja R, Messier V, D'Aoust E, Falappa CM, Justice T, Orszag A, Tschirhart H, Dallaire M, Ladouceur M, Perkins BA. Single- and Dual-Hormone Artificial Pancreas for Overnight Glucose Control in Type 1 Diabetes. J Clin Endocrinol Metab. 2016 Jan;101(1):214-23. doi: 10.1210/jc.2015-3003. Epub 2015 Nov 2. PMID 26523526